CLINICAL TRIAL: NCT06421207
Title: Open Label Study to Explore Tissue Histopathology Following Reduction in Skin Surface Using the Ellacor® Micro-Coring™ Procedure in an Abdominoplasty Model.
Brief Title: Open Label Study Exploring Tissue Histopathology After Ellacor® Procedure in an Abdominoplasty Model.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cytrellis Biosystems, Inc. (Industry)
Collaborators: Dallas Plastic Surgery Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TP-00379
Record Dates: First submitted 2024-01-29; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Histopathology; Wrinkle; Rhytides
Keywords: Mechanism of Action; Micro-Coring; Abdominoplasty; histopathology; immunohistochemistry; wrinkle treatment

STUDY DESIGN:
Intervention Model Description: Abdominoplasty model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cohort 1 Safety Evaluation of Treatment Depths (Active Comparator): Each subject will be treated a single time at 4mm, 5mm and 7 mm depths at a minimum of 3 treatment areas. A non-treated control area will also be designated. Histology evaluations for all treatment areas and the control area will occur 30 days after treatment (Day 30).
  Interventions: Device: ellacor® Micro-Coring procedure
- Cohort 2 Multiple Treatment Histology (Active Comparator): Each subject will be treated at a specified depth (4mm). Treatment area 1 will have 3 treatments with the study device, each treatment 30 days apart starting on Day 0. Treatment area 2 will have 2 treatments with the study device 30 days apart starting on Day 30. Treatment area 3 will have a single treatment with the study device on Day 60. A non-treated control area will also be designated. Histology evaluations for all treatment areas and the control area will occur 30 days after the area 3 treatment (Day 90).
  Interventions: Device: ellacor® Micro-Coring procedure

INTERVENTIONS:
Device: ellacor® Micro-Coring procedure — ellacor® Micro-Coring Technology is FDA approved for use by medical professionals for the treatment of moderate and severe wrinkles in the mid and lower face in adults aged 22 years or older with Fitzpatrick skin types I-IV.

SUMMARY:
The goal of this study to better understand how the ellacor® Micro-Coring™ procedure works using an abdominoplasty, or tummy tuck surgery, model. The people participating in the study will have already decided that they want to have an abdominoplasty procedure.

The main questions this study aims to answer are:

1. how does the ellacor® procedure change skin tissue?
2. is the ellacor® device safe to use at specific treatment depths?

The ellacor® procedure will be performed on people who are going to have abdominoplasty surgery. The ellacor® treatment areas will be limited to the areas marked for removal of skin during the abdominoplasty. The treated tissue will be sent to a lab for microscopic study after the abdominoplasty procedure is complete. A minimum of 3 people will be treated in each of 2 groups for a total of 6 total participants.

3 participants in the first group will have the ellacor® procedure done 30 days before their abdominoplasty surgery. The ellacor® procedure will be done at different depths in designated locations: 4mm, 5mm and 7mm. The participants will be asked about any changes to their health or medications while on the study.

3 participants in the second group will have the ellacor® procedure done at 3 different timepoints, 30 days apart, all at the same depth of 4mm. They will also be asked about any changes to their health or medications while on the study.

Researchers will study the abdominoplasty tissue under a microscope after it has been removed from the participants. They will compare the areas treated by the ellacor® device to an area left untreated. This will reveal any changes in the skin tissue between treated and untreated areas, if they occur.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing planned abdominoplasty
* Are willing to donate their tissue for evaluation
* BMI ≤ 30
* Women 18 years or older
* Fitzpatrick scale I-VI
* Females of childbearing potential will have a negative urine pregnancy test prior to each procedure
* Are judged to be in good health based on the results of a medical history and physical examination (standard of care for abdominoplasty) at screening
* Has been informed of the nature of the study and agrees to its provisions and has provided written informed consent on a form, as approved by the IRB of the respective clinical site.
* Able and willing to comply with all visits, procedures and evaluation schedules and requirements

Exclusion Criteria:

* Having an active bleeding disorder or currently taking anticoagulants
* History of keloid formation or abnormal wound healing
* Inflammation or active infection and treatment area
* Compromised immune system (e.g., diabetes)
* Any surgery or treatments in the abdominal area 12 months prior to procedure
* Comorbid condition that could limit ability to participate in the study or to comply with follow up requirements
* Pregnant or breastfeeding
* Tattoo and/or mole located within the planned treatment area(s)
* Vulnerable populations include those defined 45 CFR 46 Subparts B, and those mentioned in 45 CFR 46.111(b): mentally disabled persons, or economically or educationally disadvantaged persons
* Any issue that at the discretion of the investigator would contraindicate the subject's participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-representation.
Enrollment: 6 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Adverse events will be collected from Day 0 (the initial ellacor treatment day) through the day of the scheduled abdominoplasty procedure (Day 30 for Cohort 1 or Day 90 for Cohort 2).
  The incidence and severity of adverse events will be evaluated for both Study Cohorts.
The change in histopathology of abdominoplasty tissue samples after a single treatment with the ellacor® device at depths of 4mm, 5mm and 7mm as compared to an untreated control area. | Histopathological studies will be performed on excised abdominoplasty tissue approximately 30 days after a single ellacor® treatment.
  Compare histopathology of stained tissue isolated after a single ellacor® treatment on abdominal tissue. Tissue being evaluated by staining will be isolated from excised abdominal tissue following abdominoplasty. Tissue will have an untreated control area compared to three treated areas wherein the depth of treatment will be 4mm, 5mm, and 7mm. The evaluation will include staining with: Hematoxylin and Eosin (H&E), Herovici, and Movat stains. The use of these stains will provide a comparison of the structural tissue changes (H&E stain), change in the presence of Type III (young) collagen and Type I (mature) collagen (Herovici stain) and change in the presence of collagen, fibrin and elastic fibers (Movat stain) of treated areas compared to untreated control area. Histopathology of the excised abdominal tissue will be performed at a central pathology laboratory by a designated pathologist who will provide detailed report of the findings.
The change in histopathology of abdominoplasty tissue after 1, 2 and 3 ellacor® treatments (depth of 4mm) compared to untreated control area. Treatments are separated by 30 days with a final tissue comparison 90 days after the first treatment. | The histopathological studies will be performed on the excised abdominoplasty tissue approximately 90 days after the first ellacor® treatment, 60 days after the second treatment and 30 days after the final treatment is performed.
  Evaluate the comparative histopathology of tissue isolated after multiple treatments on abdominal tissue. Tissue being evaluated by staining will be isolated from excised abdominal tissue after abdominoplasty. Tissue will have an untreated control area compared to three treated areas. Area 1 will have 3 treatments. Area 2 will have 2 treatments. Area 3 will have treatment. The evaluation will include staining with: Hematoxylin and Eosin, Herovici, and Movat stains. These stains will provide comparison of the structural tissue change (H&E stain), change in the presence of Type III (young) and Type I (mature) collagen (Herovici stain) and change in the presence of collagen, fibrin and elastic fibers (Movat stain) of treated areas compared to the untreated control area. Histopathology of the excised abdominal tissue will be performed at a central pathology laboratory by a designated pathologist who will provide detailed report of the findings.

CONTACTS AND LOCATIONS:
Overall Officials: Rod Rohrich, MD, Principal Investigator — Dallas Plastic Surgery Institute
Locations (1):
- Dallas Plastic Surgery Institute, Dallas, Texas, United States